CLINICAL TRIAL: NCT04027166
Title: Effects of Methadone on Cognitive Function and Pain Threshold
Brief Title: Cognitive Function and Pain Threshold in People Who Are Methadone Maintained
Acronym: OUD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Mehmet Sofuoglu, Principal Investigator, Yale University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MS057
Record Dates: First submitted 2019-07-10; First posted 2019-07-19 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Methadone

STUDY DESIGN:
Intervention Model Description: This within-subject study design will assess pain and cognitive performance in individuals with OUD engaged in MMT. Participants will be asked to complete two separate 4 hours sessions that will be spaced approximately 2-15 days apart. The two sessions will differ based on methadone administration to evaluate study variables in methadone peak (immediately after dose) and trough (20-24 hour after last dose) states.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- administration immediate (Experimental): Methadone will be administered prior to study procedures
  Interventions: Drug: Methadone
- administration delayed (Experimental): Methadone will be held for four hours until the end of all study procedures.
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Methadone — Methadone will be administered before study procedures
  Arms: administration immediate
Drug: Methadone — Methadone will be delayed (4 hours) until the end of the procedures
  Arms: administration delayed

SUMMARY:
Male and female participants, over the age of 18, with OUD currently receiving methadone will be enrolled. This within-subject study design will assess pain and cognitive performance in individuals with OUD engaged in MMT. Participants will be asked to complete two separate 4-hour sessions that will be spaced approximately 2-15 days apart. The two sessions will differ based on methadone administration to evaluate study variables in methadone peak (immediately after dose) and trough (20-24 hour after last dose) states. The order of these sessions will be counterbalanced across participants. At the beginning of each session, participants will complete a pain sensitivity task at baseline and post-methadone administration to determine pain threshold and tolerance. Participants will then complete computerized cognitive assessments of working memory, set-shifting, attentional bias, and behavioral inhibition. The cognitive assessments will administered across three time-points (0, 90, and 180 minutes). Pain threshold and tolerance will be measured again after 240 minutes. In addition, opioid craving, withdrawal, pain intensity, and emotional valence will be repeatedly assessed during 240 minute session.

DETAILED DESCRIPTION:
After completion of the phone screen, eligible participants will be brought into the laboratory, given a description of the study, and assessed on inclusion and exclusion criteria by research personnel. Details pertaining to the cognitive measures, pain measures, and methadone manipulation will be discussed and informed consent will be obtained along with a signed release to allow study personnel to monitor opioid maintenance. Information on medical, psychiatric and drug use histories will be collected. Individuals with a history of vascular problems or high blood pressure will be evaluated by the research physician. In addition, laboratory tests collecting information on blood alcohol content and urine toxicology will be conducted. Participants will be deemed ineligible to participate if they are not medically cleared by research clinician. Veterans who have a positive BAC will be rescheduled and the methadone maintenance program's clinical protocol will be implemented.

All sessions will be conducted at the West Haven VA Connecticut Healthcare Campus. Participants will be asked to complete two sessions, approximately 2-15 days apart. Order of peak and trough sessions will be counterbalanced between participants. Each session will last approximately four hours. Prior to each testing session, participants will be asked to refrain from caffeine for at least one hour. They will be served a standardized breakfast (i.e., bagel and cream cheese) and offered one smoke break prior to beginning the experimental session. They will be asked to refrain from smoking until the completion of the study protocol. Methadone administration will be coordinated with methadone maintenance treatment staff to relay information about which condition the participant will complete on a given session. At the start of each session, participants will complete computerized cognitive assessments and self-report questionnaires. The computerized cognitive measures will repeated at hours 0, 1.5, and 3. Several state questionnaires will be administered at hours every 30 minutes. Participants will also complete a pain sensitivity measure (i.e., cold pressor task) to assess baseline threshold and tolerance at hour 0 and hour 4.

This study is complete with 27 enrolled and 20 completers.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, over the age of 18
* Diagnosed with opioid dependence and currently enrolled in methadone maintenance treatment
* Compliant in opioid maintenance treatment and on a stable dose for two weeks or greater
* No current medical problems deemed contraindicated for participation by physician investigator

Exclusion Criteria:

* History of psychosis as determined by review of EMR.
* Acute suicidal ideation.
* History of medical conditions that the physician investigator deems contraindicated for inclusion in the study (e.g., untreated hypertension)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
changes in cognitive functioning using the go no go task | up to 24 months
  during methadone peak and trough states.

SECONDARY OUTCOMES:
self-reported measures of pain from the cold pressor test | up to 24 months
  during methadone peak and trough states

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sofuoglu, M.D., Ph.D., Principal Investigator — Veteran Affairs Hospital
Locations (1):
- Veteran Affairs Hospital, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be de-identified and will only be used with this Principle Investigator.